CLINICAL TRIAL: NCT00250679
Title: Multicenter, Double-Blind, Double-Dummy, Randomized, Active-Controlled, Parallel Group Long-Term Safety Study of 15 μg and 25 μg Arformoterol Tartrate Inhalation Solution BID in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Safety and Efficacy of Arformoterol Tartrate Inhalation Solution in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 091-061
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Results first posted 2009-02-19 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Bronchitis; Emphysema
Keywords: COPD; chronic bronchitis; emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema; Bronchitis, Chronic | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Formoterol 12 ųg 2x/day (Active Comparator)
  Interventions: Drug: Formoterol 12 ųg BID; Drug: Placebo
- Arformoterol 15 ųg 2x/day (Experimental)
  Interventions: Drug: Arformoterol tartrate inhalation solution; Drug: Placebo
- Arformoterol 25 ųg 2x/day (Experimental)
  Interventions: Drug: Arformoterol 25 ųg BID; Drug: Placebo

INTERVENTIONS:
Drug: Arformoterol tartrate inhalation solution — Arformoterol 15 ųg BID by nebulization
  Other Names: Brovana®
  Arms: Arformoterol 15 ųg 2x/day
Drug: Arformoterol 25 ųg BID — Arformoterol 25 ųg BID by nebulization
  Other Names: Brovana; R,R formoterol
  Arms: Arformoterol 25 ųg 2x/day
Drug: Formoterol 12 ųg BID — Formoterol fumarate 12 ųg BID via aerolizer/DPI
  Other Names: Foradil; R,S-formoterol
  Arms: Formoterol 12 ųg 2x/day
Drug: Placebo — Placebo nebule or placebo aerolizer

SUMMARY:
To evaluate the long-term safety and monitor the long-term efficacy of arformoterol over a period of 6 months in subjects with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This is a double-blind, double-dummy, multicenter, randomized, active-controlled, parallel group, outpatient, safety study to evaluate the long term safety of arformoterol in the treatment of subjects with COPD. Study participation will be over approximately 6 months. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects must be at least 35 years old at the time of consent
* Subjects must have a pre-established, documented primary clinical diagnosis of non-asthmatic COPD or are referred for diagnosis of non-asthmatic COPD
* Subjects must have a >=15 pack-year smoking history and a baseline breathlessness severity grade of >=2 (Modified Medical Research Council [MMRC] Dyspnea Scale Score) at Visits 1 and 2
* Female subjects <=65 years of age must have a negative serum pregnancy test, females of childbearing potential must be using an acceptable method of birth control
* Subjects must be in general good health.

Key Exclusion criteria:

* Subjects with a history of asthma, with the exception of asthma diagnosed in childhood
* Subjects with a blood eosinophil count >5% of total white blood cell count
* Subjects have had a febrile illness within 72 hours (3 days) before Screening Visit 1
* Subjects with a chest x-ray that suggests a diagnosis other than COPD (e.g., diagnostic of pneumonia, other infection, atelectasis, or pneumothorax or other active/ongoing pulmonary conditions)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sepracor Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (59):
- United States (59):
  - Birmingham, Alabama
  - Jasper, Alabama
  - Mobile, Alabama
  - Little Rock, Arkansas
  - Carmichael, California
  - Fullerton, California
  - Long Beach, California
  - Paramount, California
  - Rancho Mirage, California
  - San Diego, California
  - Walnut Creek, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Bay Pines, Florida
  - Brandon, Florida
  - Gainesville, Florida
  - Panama City, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Normal, Illinois
  - Evansville, Indiana
  - Topeka, Kansas
  - East Slidell, Louisiana
  - Lafayette, Louisiana
  - Metairie, Louisiana
  - Sunset, Louisiana
  - Baltimore, Maryland
  - Chester, Maryland
  - Wheaton, Maryland
  - Ann Arbor, Michigan
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Lake Oswego, Oregon
  - Medford, Oregon
  - Pittsburgh, Pennsylvania
  - Swarthmore, Pennsylvania
  - East Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Union, South Carolina
  - Knoxville, Tennessee
  - Houston, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Danville, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Morgantown, West Virginia

REFERENCES:
- [Background] Hanania NA, Donohue JF, Nelson H, Sciarappa K, Goodwin E, Baumgartner RA, Hanrahan JP. The safety and efficacy of arformoterol and formoterol in COPD. COPD. 2010 Feb;7(1):17-31. doi: 10.3109/15412550903499498. PMID 20214460

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients were each issued two randomization numbers; both subjects are included only once in the intent-to-treat (ITT) population. One additional subject was randomized in error and did not receive study drug. This subject is excluded from the ITT population.
Period: Overall Study
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Started | 147 | 149 | 147
Completed | 108 | 100 | 103
Not Completed | 39 | 49 | 44
Not completed — Adverse Event | 12 | 15 | 16
Not completed — Protocol Violation | 2 | 4 | 3
Not completed — Withdrawal by Subject | 15 | 18 | 15
Not completed — Lost to Follow-up | 3 | 4 | 2
Not completed — Does Not Meet Entry Criteria | 1 | 4 | 2
Not completed — Lack of Efficacy | 0 | 1 | 3
Not completed — Technical Holter issues | 1 | 0 | 2
Not completed — Moved | 1 | 1 | 0
Not completed — Non-compliance | 1 | 1 | 0
Not completed — various single events: hip surgery,diary | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day | Total
Number analyzed (Participants) | 147 | 149 | 147 | 443
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 77 | 71 | 77 | 225
  >=65 years | 70 | 78 | 70 | 218
Age Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.8) | 65.4 (9.0) | 63.8 (8.6) | 64.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 52 | 56 | 172
  Male | 83 | 97 | 91 | 271
Region of Enrollment [Number; unit: participants]
  United States | 147 | 149 | 147 | 443
# Chronic Obstructive Pulmonary Disease (COPD) Exacerbations in 30 days prior to screening [Number; unit: participants] — Number of patients with a specified number of COPD exacerbations in the 30 days prior to screening. COPD stands for 'chronic obstructive pulmonary disease' and is a progressive disease that makes it hard to breath. Exacerbations refers to a worsening of the condition.
  participants
    0 exacerbations | 146 | 147 | 145 | 438
    1 exacerbation | 1 | 2 | 1 | 4
    2 exacerbations | 0 | 0 | 0 | 0
    >2 exacerbations | 0 | 0 | 1 | 1
# Packs Currently Smoked Per Day [Number; unit: participants] — Number of participants with a specified range of packs of cigarettes smoked per day.
  participants
    0 packs per day | 72 | 89 | 82 | 243
    >0 - <=1 packs per day | 59 | 38 | 44 | 141
    >1 - <=2 packs per day | 14 | 21 | 17 | 52
    >2 - <=4 packs per day | 2 | 1 | 4 | 7
    >4 packs per day | 0 | 0 | 0 | 0
Number of Pack-Years Smoked [Number; unit: participants] — Number of participants with a specified number range of pack years smoked. Number of pack years smoked is defined as the number of cigarette packs smoked per day times the number of years smoked.
  participants
    < 15 pack years smoked | 0 | 0 | 0 | 0
    >= 15 - < 25 pack years smoked | 8 | 13 | 13 | 34
    >= 25 - < 30 pack years smoked | 10 | 10 | 11 | 31
    >= 30 pack years smoked | 129 | 126 | 123 | 378
Oral or Inhaled Steroid Use [Number; unit: participants] — Number of participants taking oral or inhaled corticosteriod at baseline. These were allowed at study entry and for the duration of the study as long as the regimen was stable for at least 14 days prior to entry and throughout the study.
  participants
    Yes | 52 | 59 | 59 | 170
    No | 95 | 90 | 88 | 273
Race/Ethnicity [Number; unit: participants]
  Asian | 0 | 0 | 0 | 0
  Black or African American | 19 | 21 | 23 | 63
  Caucasian | 127 | 126 | 122 | 375
  Hispanic | 1 | 1 | 2 | 4
  Other | 0 | 1 | 0 | 1
Baseline Dyspnea Index [Mean (Standard Deviation); unit: units on a scale] — Baseline Dyspnea Index (range 0-12) is defined to be the sum of the Functional Impairment, Magnitude of Task, and Magnitude of Effort scores (each on a 0-4 scale) obtained at visit 2 (baseline). On each scale, a high measurement represents the most impairment to health.
  units on a scale | 5.34 (1.72) | 5.34 (2.18) | 5.10 (2.38) | 5.26 (2.09)
Forced Expiratory Volume (FEV1) [Mean (Standard Deviation); unit: Liter] — FEV1 stands for 'forced expiratory volume 1 second'. It is the amount of air that you can forcibly blow out in one second, measured in liters
  Liter | 1.210 (0.420) | 1.222 (0.465) | 1.204 (0.422) | 1.212 (0.435)
Percent Predicted Forced Expiratory Volume (FEV1) [Mean (Standard Deviation); unit: percent predicted FEV1] — FEV1 stands for 'forced expiratory volume 1 second'. It is the amount of air that you can forcibly blow out in one second, measured in liters. FEV1 can be predicted using patients' height and age. This value is the percent of the predicted FEV1.
  percent predicted FEV1 | 41.19 (11.52) | 40.87 (13.59) | 40.22 (12.22) | 40.76 (12.46)

OUTCOME MEASURES:

1. Primary Outcome: Percent (%) of Participants With Adverse Events (AEs), in Particular COPD Exacerbations
Description: Percent of participants with the adverse event specified.
  SOC = system organ class.
Time Frame: Six months
Population: ITT Population
Measure: Number; unit: percent of participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
percent of participants
  Any AE | 66.7 | 67.8 | 76.2
  Any Severe AE | 10.9 | 13.4 | 11.6
  Any Potentially Related AE | 34.7 | 32.9 | 34.7
  Any Beta-Mediated AE | 17.0 | 10.7 | 15.6
  Any AE w SOC of Cardiac Disorders | 6.1 | 6.0 | 6.1
  Any Serious AE | 9.5 | 13.4 | 6.8
  Any AE Leading to Discontinuation | 8.2 | 10.1 | 12.2
  Any COPD Exacerbation (Protocol Definition) | 22.4 | 32.2 | 30.6
  Any COPD Exacerbation (Expanded Definition) | 27.9 | 35.6 | 38.1
  Any Ischaemic AE | 1.4 | 0.7 | 5.4
  Any Arrhythmnic AE | 3.4 | 3.4 | 1.4
  Any AE w SOC Respiratory, Thoracic, & Mediastinal | 27.2 | 34.2 | 34.0

2. Secondary Outcome: Number of Participants With New 24-Hour Holter Monitoring Alerts
Description: New holter monitoring alerts are defined as those alerts that occurred post-randomization and were not present at baseline.
Time Frame: Visit 6 (week 27)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Participants | 15 | 19 | 9

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Glucose Evaluations
Description: Patients with glucose values that met low (<=40 mg/dL) or high (>=175 mg/dL) criteria were considered potentially clinically significant.
Time Frame: visit 6 (week 27)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Participants
  <=40 mg/dL | 1 | 0 | 1
  >=175 mg/dL | 20 | 55 | 54

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Potassium Evaluations
Description: Patients with potassium values that met low (<=3 mEq/L) or high (>=6 mEq/L) criteria were considered potentially clinically significant.
Time Frame: visit 6 (week 27)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Participants
  <= 3mEq/L | 2 | 4 | 3
  >= 6mEq/L | 4 | 1 | 1

5. Secondary Outcome: Number of Participants With New 12-Lead Electrocardiogram (ECG) Alerts
Description: New Electrocardiogram (ECG) alerts are defined as those alerts that occurred post-treatment and were not present at baseline.
Time Frame: visit 6 (week 27)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Participants | 1 | 1 | 5

6. Secondary Outcome: Inspiratory Capacity Changes From Baseline
Description: Mean Change in Inspiratory Capacity values from baseline (baseline assessment obtained at Visit 2, pre-dose). Spirometry measurements collected within 6 hours following in-clinic rescue/supplemental medications use were excluded from analysis.
Time Frame: weeks 0,3,13,26
Population: ITT Population This outcome was added as an amendment after the study was initiated; therefore approximately half of the ITT population had these assessments at baseline. An available cases analysis was performed with no imputation for missing data.
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Liter
  Visit 2 (wk 0): 2 hours Post-dose n=79,85,80 | 0.240 (0.363) [0.158 to 0.321] | 0.297 (0.300) [0.232 to 0.361] | 0.330 (0.354) [0.251 to 0.408]
  Visit 3 (wk 3): Pre-Dose n=74,77,69 | 0.058 (0.380) [-0.030 to 0.146] | 0.032 (0.409) [-0.060 to 0.125] | 0.124 (0.370) [0.035 to 0.212]
  Visit 3 (wk 3): 2 hours Post-dose n=75,75,69 | 0.206 (0.410) [0.111 to 0.300] | 0.241 (0.401) [0.149 to 0.333] | 0.331 (0.448) [0.223 to 0.438]
  Visit 4 (wk 13): Pre-Dose n=62,63,58 | 0.114 (0.368) [0.020 to 0.207] | 0.005 (0.441) [-0.106 to 0.116] | 0.124 (0.447) [0.006 to 0.242]
  Visit 4 (wk 13): 2 hours Post-Dose n=60,63,58 | 0.290 (0.445) [0.174 to 0.405] | 0.233 (0.364) [0.141 to 0.325] | 0.284 (0.423) [0.173 to 0.395]
  Visit 5 (wk 26): Pre-Dose n=58,58,53 | 0.039 (0.354) [-0.054 to 0.132] | 0.057 (0.326) [-0.029 to 0.142] | 0.154 (0.371) [0.051 to 0.256]
  Visit 5 (wk 26): 2 hours Post-Dose n=58,58,53 | 0.234 (0.451) [0.116 to 0.353] | 0.202 (0.402) [0.097 to 0.308] | 0.368 (0.443) [0.245 to 0.490]

7. Secondary Outcome: 6-Hour Peak Changes From Baseline in Forced Expiratory Volume (FEV1)
Description: The 6 hour peak change from baseline is the maximum of the post-dose change values through 6 hours at each visit.
Time Frame: weeks 0,3,13,26
Population: ITT population. An available cases analysis was performed with no imputation for missing data.
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Liter
  Visit 2 (week 0) n=147,149,147 | 0.294 (0.210) [0.260 to 0.328] | 0.314 (0.189) [0.284 to 0.345] | 0.357 (0.218) [0.321 to 0.392]
  Visit 3 (week 3) n=133,133,131 | 0.280 (0.229) [0.241 to 0.319] | 0.305 (0.211) [0.269 to 0.341] | 0.334 (0.230) [0.294 to 0.374]
  Visit 4 (week 13) n=117,112,111 | 0.251 (0.223) [0.210 to 0.291] | 0.316 (0.236) [0.271 to 0.360] | 0.323 (0.222) [0.281 to 0.365]
  Visit 5 (week 26) n=108,100,103 | 0.264 (0.230) [0.220 to 0.308] | 0.302 (0.239) [0.255 to 0.349] | 0.343 (0.224) [0.299 to 0.387]

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Heart Rate
Description: Number of subjects with a heart rate that was lower/higher than a set limit and increased/decreased from set baseline limit in beats per minute (bpm)
Time Frame: visit 6 (week 27)
Measure: Number; unit: Participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Participants
  < 50 bpm & >= 15 bpm | 6 | 5 | 2
  < 120 bpm & >= 25 bpm | 2 | 1 | 1

9. Secondary Outcome: Ipratropium Bromide Metered Dose Inhaler (MDI) Usage: Days Used Per Week
Description: Supplemental medication usage is recorded throughout the study. MDI stands for metered dose inhaler.
Time Frame: Screening (day-14 to 0) and Treatment (week 0 - 26)
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: Days Used / Week
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Days Used / Week
  Screening Period (day -14 to day 0 pre-dose) | 4.10 (2.92) [3.62 to 4.57] | 3.73 (2.95) [3.25 to 4.21] | 3.84 (2.92) [3.36 to 4.31]
  Visits 2-5 (week 0 - 26) | 2.66 (2.63) [2.33 to 3.09] | 2.36 (2.60) [1.94 to 2.78] | 2.52 (2.66) [2.09 to 2.96]

10. Secondary Outcome: Ipratropium Bromide Metered Dose Inhaler (MDI) Usage: Number of Actuations Per Day
Description: Supplemental medication usage during the study. MDI stands for metered dose inhaler. An actuation is one depression of the device that releases medication.
Time Frame: Screening (day-14 to 0) and Treatment (week 0 - 26)
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: Actuations / Day
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Actuations / Day
  Screening period (day -14 to day 0 pre-dose) | 2.70 (2.72) [2.25 to 3.14] | 2.43 (2.69) [1.99 to 2.86] | 2.67 (3.06) [2.18 to 3.17]
  Visits 2-5 (week 0 - 26) | 1.61 (2.28) [1.24 to 1.98] | 1.59 (2.37) [1.21 to 1.97] | 1.58 (2.12) [1.24 to 1.93]

11. Secondary Outcome: Racemic Albuterol or Levalbuterol Metered Dose Inhaler (MDI) Usage: Days Used Per Week
Description: Rescue medication usage during the study. MDI stands for metered dose inhaler.
Time Frame: Screening (day-14 to 0) and Treatment (week 0 - 26)
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: Days Used / Week
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Days Used / Week
  Screening Period (day -14 to day 0 pre-dose) | 4.18 (2.85) [3.72 to 4.65] | 4.20 (2.86) [3.74 to 4.66] | 4.23 (2.77) [3.78 to 4.69]
  Visits 2-5 (week 0 - 26) | 2.85 (2.64) [2.42 to 3.28] | 2.44 (2.49) [2.03 to 2.84] | 2.75 (2.64) [2.32 to 3.18]

12. Secondary Outcome: Racemic Albuterol or Levalbuterol Metered Dose Inhaler (MDI) Usage: Number of Actuations Per Day
Description: Rescue medication usage during the study. MDI stands for metered dose inhaler. An actuation is one depression of the device that releases medication.
Time Frame: Screening (day-14 to 0) and Treatment (week 0 - 26)
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: Actuations/Day
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Actuations/Day
  Screening Period (day -14 to day 0 pre-dose) | 2.91 (2.80) [2.45 to 3.37] | 2.68 (2.57) [2.27 to 3.10] | 2.97 (3.05) [2.47 to 3.47]
  Visits 2-5 (week 0 - 26) | 1.71 (2.27) [1.34 to 2.08] | 1.56 (2.32) [1.18 to 1.93] | 1.65 (2.11) [1.31 to 2.00]

13. Secondary Outcome: Time-Normalized Area Under the Curve (nAUC) From 0 to 6 Hrs for Forced Expiratory Volume in One Second (FEV1) Changes From Baseline
Description: Area under the change from baseline curve from 0 to 6 hours. Time-normalized AUC (0-6 hrs) was derived using the linear trapezoidal method.
Time Frame: weeks 0,3,13,26
Population: ITT Population. Spirometry measurements collected within 6 hours following in-clinic rescue/supplemental medications use were excluded from analysis.
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Liter
  Visit 2 (week 0) n=147,149,147 | 0.191 (0.172) [0.163 to 0.219] | 0.216 (0.157) [0.191 to 0.242] | 0.253 (0.179) [0.224 to 0.282]
  Visit 3 (week 3) n=129,129,131 | 0.175 (0.204) [0.139 to 0.210] | 0.208 (0.200) [0.173 to 0.243] | 0.224 (0.206) [0.188 to 0.259]
  Visit 4 (week 13) n=113,110,110 | 0.155 (0.210) [0.116 to 0.194] | 0.214 (0.225) [0.171 to 0.256] | 0.218 (0.214) [0.177 to 0.258]
  Visit 5 (week 26) n=107,100,101 | 0.161 (0.209) [0.121 to 0.201] | 0.197 (0.229) [0.152 to 0.243] | 0.241 (0.209) [0.200 to 0.282]

14. Secondary Outcome: Transitional (Relative Change in) Dyspnea Index
Description: The transitional focal score (-9 to 9) is the sum of relative change from baseline for the Functional Impairment, Magnitude of Task, and Magnitude of Effort scores (each -3 to 3 scale). A Transitional Dyspnea Index score of -9 represents a maximum degradation of all three tests; a score of 9 represents a maximum improvement of all three tests.
Time Frame: weeks 13, 26
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 4 (week 13) n=115,113,114 | 1.50 (2.40) [1.05 to 1.94] | 1.47 (2.56) [0.99 to 1.95] | 1.56 (2.74) [1.05 to 2.07]
  Visit 5 (week 26) n=108,102,103 | 1.44 (2.77) [0.92 to 1.97] | 1.43 (2.83) [0.88 to 1.99] | 1.49 (2.76) [0.95 to 2.02]

15. Secondary Outcome: Number of Participants With an Improved Transitional Dyspnea Index
Description: The number of participants with a transitional focal score (range -9 to 9) of >=1 improvement. Transitional focal score compares current health against baseline for the Functional Impairment, Magnitude of Task, and Magnitude of Effort scores. A score of -9 is maximum worsening and 9 is maximum improvement.
Time Frame: weeks 13, 26
Population: ITT Population. Visit 4 n=115,113,114 Visit 5 n=108,102,103
Measure: Number; unit: Participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Participants
  >= 1Unit Improvement, visit 4 (wk13) n=115,113,114 | 59 | 59 | 61
  >= 1 Unit Improvement,visit 5(wk 26) n=108,102,103 | 56 | 49 | 54

16. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Changes From Baseline for 24 Hour Post Dose Timepoint (Trough)
Description: The 24 hour trough is the FEV1 value obtained 24 hours post first dose. This value is compared to the baseline FEV1 value.
Time Frame: weeks 0,3,13,26
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Liters
  Visit 2 (week 0) n=141,143,141 | 0.162 (0.209) [0.127 to 0.197] | 0.172 (0.206) [0.138 to 0.206] | 0.155 (0.226) [0.117 to 0.192]
  Visit 3 (week 3) n=130,130,127 | 0.096 (0.192) [0.063 to 0.130] | 0.124 (0.209) [0.088 to 0.161] | 0.131 (0.201) [0.096 to 0.167]
  Visit 4 (week 13) n=111,108,110 | 0.094 (0.192) [0.058 to 0.130] | 0.116 (0.187) [0.080 to 0.152] | 0.101 (0.207) [0.062 to 0.140]
  Visit 5 (week 26) n=105,97,101 | 0.087 (0.215) [0.046 to 0.129] | 0.098 (0.243) [0.049 to 0.147] | 0.137 (0.229) [0.091 to 0.182]

17. Secondary Outcome: Subject Global Evaluations Change From Baseline
Description: The global evaluation is a COPD symptoms rating ranging from 1 to 7, with 1=much better and 7=much worse. Ratings were assessed relative to the subject's initial entry into the study.
Time Frame: weeks 13, 26
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 4 (week 13) n=112,112,114 | -0.96 (1.39) [-1.23 to -0.70] | -1.11 (1.51) [-1.39 to -0.82] | -0.89 (1.49) [-1.16 to -0.61]
  Visit 5 (week 26) n=106,102,102 | -0.97 (1.50) [-1.26 to -0.68] | -1.06 (1.41) [-1.33 to -0.78] | -0.83 (1.70) [-1.17 to -0.50]

18. Secondary Outcome: Investigator Global Evaluations Change From Baseline
Description: The global evaluation is a COPD symptoms rating ranging from 1 to 7, with 1 = much better and 7 = much worse. Ratings were assessed relative to the subject's initial entry into the study.
Time Frame: weeks 13, 26
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 4 (week 13) n=111,112,110 | -0.66 (1.27) [-0.90 to -0.42] | -0.88 (1.27) [-1.11 to -0.64] | -0.75 (1.43) [-1.02 to -0.48]
  Visit 5 (week 26) n=106,100,100 | -0.74 (1.20) [-0.97 to -0.51] | -0.74 (1.28) [-0.99 to -0.49] | -0.76 (1.65) [-1.09 to -0.43]

19. Secondary Outcome: BODE Index
Description: The BODE index (0=relative health and 10=severe chronic obstructive pulmonary disease) is a multi-dimension COPD grading system that incorporates body-mass index (B), degree of airflow obstruction (O), dyspnea (D), and exercise capacity (E) as measured by the 6-minute walk test. Scores were derived using pre-dose assessments from each visit.
Time Frame: Baseline (visit 2), weeks 13, 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 2 (baseline- week 0) n=146,148,147 | 4.82 (1.58) | 4.98 (1.64) | 5.14 (1.73)
  Visit 4 (week 13) n=110,108,109 | 4.22 (2.03) | 3.97 (1.90) | 4.28 (1.95)
  Visit 5 (week 26) n=103,100,101 | 3.92 (1.91) | 3.94 (1.99) | 4.11 (2.20)

20. Secondary Outcome: 6-Minute Walk: Change From Baseline in the Distance Walked in 6 Minutes
Description: Mean change from baseline in distance walked (meters)
Time Frame: Post-Dose weeks 0, 13, 26
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
meters
  Visit 2 (week 0 - post dose) n=146,148,146 | 15.28 (81.22) [2.00 to 28.56] | 15.72 (67.59) [4.74 to 26.70] | 12.37 (69.65) [0.97 to 23.76]
  Visit 4 (week 13 - post dose) n=116,110,112 | 16.05 (104.90) [-3.24 to 35.34] | 4.13 (128.01) [-20.06 to 28.32] | 31.07 (77.20) [16.61 to 45.52]
  Visit 5 (week 26 - post dose) n=106,97,103 | 24.42 (94.19) [6.28 to 42.56] | 1.24 (135.05) [-25.98 to 28.46] | 37.00 (85.01) [20.38 to 53.61]

21. Secondary Outcome: Mean Change From Baseline in St. George's Respiratory Questionnaire
Description: Scores are expressed as a mean change from baseline of overall impairment (total score). The questionnaire has a scale of 100 which represents worst possible health status to 0 which indicates best possible health status.
Time Frame: weeks 13, 26
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 4 (week 13) n=105,102,105 | -4.16 (10.09) [-6.11 to -2.21] | -3.44 (12.10) [-5.81 to -1.06] | -1.92 (9.86) [-3.82 to -0.01]
  Visit 5 (week 26) n=97,94,97 | -6.76 (10.06) [-8.78 to -4.73] | -3.73 (13.14) [-6.42 to -1.04] | -3.68 (11.78) [-6.06 to -1.31]

22. Secondary Outcome: Number of Participants With a >=4 Unit Improvement on the St. George's Respiratory Questionnaire
Description: Scores are expressed as the number of participants with >= 4 unit improvement in overall impairment (total score), where 100 represents worst possible health status and 0 indicates best possible health status.
Time Frame: Visit 4 (week 13) , Visit 5 (week 26)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Participants
  Visit 4 (week 13) n=105,102,105 | 49 | 47 | 39
  Visit 5 (week 26) n=97,94,97 | 55 | 43 | 42

23. Secondary Outcome: Modified Medical Research Council Dyspnea Questionaire
Description: Scores range from 0 to 4, with a score of 4 indicating that a subject is too breathless to leave the house or becomes breathless when dressing or undressing. The highest numbered question to which the subject answered 'Yes' is the Dyspnea Scale Score.
Time Frame: Baseline (visit 2), weeks 13, 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Baseline (visit 2, week 0) n=147,149,145 | 2.73 (0.78) | 2.76 (0.79) | 2.91 (0.81)
  Visit 3 (week 3) n=132,131,128 | 2.33 (1.02) | 2.47 (0.96) | 2.50 (1.12)
  Visit 4 (week 13) n=117,113,115 | 2.35 (1.03) | 2.10 (1.05) | 2.43 (1.21)
  Visit 5 (week 26) n=107,103,103 | 2.16 (1.10) | 2.09 (1.14) | 2.26 (1.26)

24. Secondary Outcome: Percent (%) of Participants With an Improved Transitional Dyspnea Index
Description: The percentage of participants with a transitional focal score (range -9 to 9) of >=1 improvement. Transitional focal score is the sum of the Functional Impairment, Magnitude of Task, and Magnitude of Effort scores. A score of -9 is maximum worsening and 9 is maximum improvement.
Time Frame: visits 4 (week 13), visit 5 (week 26)
Population: ITT population. Percentages were based on the number of subjects with non-missing data.
  Visit 4 n=115, 113, 114 Visit 5 n=108, 102, 103
Measure: Number; unit: percent of participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
percent of participants
  >=1 Unit Improvement,visit 4 (wk 13) n=115,113,114 | 51.3 | 52.2 | 53.5
  >=1 Unit Improvement,visit 5 (wk 26) n=108,102,103 | 51.9 | 48.0 | 52.4

25. Secondary Outcome: Percent (%) of Participants With a >=4 Unit Improvement in the St. George's Respiratory Questionaire
Description: Percent of participants with a >=4 unit improvement in the overall impairment (total score) of the St. George's Respiratory Questionaire. This questionaire uses a 100 - 0 scale, where 100 represents the worst possible health status and 0 indicates the best possible health status.
Time Frame: visit 4 (week 13), visit 5 (week 26)
Population: ITT population
Measure: Number; unit: percent of participants
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
percent of participants
  Visit 4 (week 13), n=105,102,105 | 46.7 | 46.1 | 37.1
  Visit 5 (week 26), n=97,94,97 | 56.7 | 45.7 | 43.3

26. Secondary Outcome: Mean Values for the 6-Minute Walk Test: Distance Walked in Meters
Description: This test measures the participants' level of fitness. It is a measure of the distance the participant can walk in 6 minutes.
Time Frame: Baseline (Visit 2), week 13, week 26
Population: ITT population
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
meters
  Visit 2 (week 0) Pre-Dose n=147, 148, 147 | 334.84 (155.43) | 315.94 (131.74) | 328.36 (183.44)
  Visit 2 (week 0) Post-Dose n=146, 149, 146 | 352.19 (163.27) | 332.80 (135.79) | 339.81 (194.09)
  Visit 4 (week 13) Pre-Dose n=115, 111, 111 | 344.95 (175.53) | 332.25 (140.60) | 333.63 (150.55)
  Visit 4 (week 13) Post-Dose n=116, 111, 112 | 352.51 (167.90) | 337.28 (165.02) | 337.68 (155.65)
  Visit 5 (week 26) Pre-Dose n=105, 100, 103 | 355.83 (181.84) | 338.21 (129.68) | 337.25 (167.83)
  Visit 5 (week 26) Post-Dose n=106, 98, 103 | 361.72 (169.96) | 344.98 (122.38) | 348.11 (174.38)

27. Secondary Outcome: Mean Values for Investigator Global Evaluations
Description: The investigator global evaluation is reported by the study investigator. It is a COPD symptoms rating ranging from 1 to 7, with 1 = much better and 7 = much worse.
Time Frame: Baseline (Visit 2), Weeks 13, 26
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 2 (Baseline, Week 0) n=145,148,144 | 3.73 (0.88) | 3.88 (0.77) | 3.84 (1.06)
  Visit 4 (week 13) n=113,112,112 | 3.12 (1.05) | 3.04 (1.17) | 3.04 (1.14)
  Visit 5 (week 26) n=107,100,102 | 3.08 (1.04) | 3.16 (1.28) | 3.01 (1.16)

28. Secondary Outcome: Mean Values for St. George's Respiratory Questionnaire
Description: A questionnaire to assess respiratory health. Scores are expressed as a percentage of overall impairment (total score), where 100 represents the worst possible health status and 0 indicates best possible health status.
Time Frame: Baseline (Visit 2), weeks 13, 26
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 2 (Baseline; week 0) n=136,141,144 | 48.86 (14.90) | 49.36 (17.38) | 52.40 (17.71)
  Visit 4 (week 13) n=114, 105, 108 | 43.48 (16.53) | 43.64 (18.94) | 49.95 (19.67)
  Visit 5 (week 26) n=105, 97, 99 | 41.72 (16.35) | 42.69 (17.98) | 48.09 (20.68)

29. Secondary Outcome: Mean Values for Subject Global Evaluations
Description: The subject global evaluation is reported by study subjects/participants. It is a COPD symptoms rating ranging from 1 to 7, with 1 = much better and 7 = much worse.
Time Frame: Baseline (Visit 2), weeks 13, 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
units on a scale
  Visit 2 (baseline; week 0) n=145, 148, 146 | 3.73 (1.08) | 3.97 (1.08) | 3.86 (1.05)
  Visit 4 (week 13) n=114, 113, 115 | 2.83 (1.09) | 2.88 (1.26) | 2.94 (1.32)
  Visit 5 (week 26) n=108, 103, 103 | 2.86 (1.31) | 2.96 (1.32) | 2.94 (1.36)

30. Secondary Outcome: Mean Values for Inspiratory Capacity
Description: Inspiratory capacity is the maximum volume that can be inhaled.
Time Frame: Baseline (Visit 2), Weeks 3, 13, 26
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Liters
  Visit 2 (wk 0, baseline) pre-dose; n=80,86,82 | 1.739 (0.630) | 1.864 (0.551) | 1.764 (0.577)
  Visit 3 (wk 3) pre-dose; n=81,83,74 | 1.826 (0.654) | 1.889 (0.558) | 1.909 (0.633)
  Visit 4 (wk 13) pre-dose; n=100,94,99 | 1.874 (0.676) | 1.890 (0.656) | 1.962 (0.640)
  Visit 5 (wk 26) pre-dose; n=106,101,101 | 1.817 (0.620) | 1.901 (0.630) | 2.070 (0.691)
  Visit 2 (wk 0, baseline) post dose; n=80,85,81 | 1.976 (0.730) | 2.161 (0.624) | 2.109 (0.610)
  VIsit 3 (wk 3) post dose; n=82,81,74 | 1.973 (0.685) | 2.111 (0.627) | 2.108 (0.632)
  Visit 4 (wk 13) post dose; n=98,94,99 | 2.089 (0.729) | 2.081 (0.658) | 2.176 (0.692)
  Visit 5 (wk 26) post dose; n=105,100,101 | 1.978 (0.690) | 2.084 (0.613) | 2.273 (0.692)

31. Secondary Outcome: Mean Values for Forced Expiratory Volume in One Second (FEV1)
Description: Forced Expiratory Volume in one second
Time Frame: Baseline (Visit 2), weeks 3, 13, 26
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Number analyzed (Participants) | 147 | 149 | 147
Liters
  Visit 2 (wk 0, baseline) pre dose; n=147,149,147 | 1.210 (0.420) | 1.222 (0.465) | 1.204 (0.422)
  Visit 2 (wk 0) 24 hr; n=141,143,141 | 1.378 (0.497) | 1.400 (0.545) | 1.360 (0.470)
  Visit 3 (wk 3) pre dose; n=129,129,132 | 1.311 (0.458) | 1.323 (0.484) | 1.327 (0.477)
  Visit 3 (wk 3) 24 hr; n=130,130,127 | 1.310 (0.456) | 1.346 (0.490) | 1.355 (0.475)
  Visit 4 (wk 13) pre dose; n=113,111,111 | 1.281 (0.470) | 1.310 (0.483) | 1.308 (0.473)
  Visit 4 (wk 13) 24 hr; n=111,108,110 | 1.316 (0.461) | 1.331 (0.460) | 1.294 (0.444)
  Visit 5 (wk 26) pre dose; n=107,102,101 | 1.283 (0.466) | 1.291 (0.453) | 1.325 (0.451)
  Visit 5 (wk 26) 24 hr; n=105,97,101 | 1.296 (0.455) | 1.314 (0.467) | 1.360 (0.468)
  Visit 2 (wk 0) 6 hr; n=142,145,138 | 1.383 (0.511) | 1.410 (0.533) | 1.428 (0.479)
  Visit 3 (wk 3) 6 hr; n=130,125,127 | 1.338 (0.464) | 1.386 (0.504) | 1.386 (0.484)
  Visit 4 (wk 13) 6 hr; n=109,109,104 | 1.339 (0.487) | 1.385 (0.482) | 1.361 (0.463)
  Visti 5 (wk 26) 6 hr; n=101,95,101 | 1.310 (0.475) | 1.355 (0.457) | 1.384 (0.483)

ADVERSE EVENTS:
Arm/Group | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Serious Adverse Events (participants affected / at risk) | 14 | 20 | 10
Other Adverse Events (participants affected / at risk) | 96 | 97 | 109
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Acute coronary syndrome (Cardiac disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Acute myocardial infarction (Cardiac disorders) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Angina pectoris (Cardiac disorders) | 1/147 (1) | 0/149 (0) | 0/147 (0)
Angina unstable (Cardiac disorders) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Atrial fibrillation (Cardiac disorders) | 1/147 (1) | 1/149 (1) | 1/147 (1)
Atrial flutter (Cardiac disorders) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Cardiac failure congestive (Cardiac disorders) | 0/147 (0) | 2/149 (2) | 1/147 (1)
Coronary artery disease (Cardiac disorders) | 1/147 (1) | 0/149 (0) | 0/147 (0)
Coronary artery thrombosis (Cardiac disorders) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Myocardial infarction (Cardiac disorders) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Supraventricular tachycardia (Cardiac disorders) | 1/147 (1) | 0/149 (0) | 0/147 (0)
Abdominal hernia (Gastrointestinal disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1/147 (1) | 0/149 (0) | 0/147 (0)
Peritonitis (Gastrointestinal disorders) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Umbilical hernia (Gastrointestinal disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Appendicitis (Infections and infestations) | 0/147 (0) | 1/149 (1) | 1/147 (1)
Gasteroenteritis viral (Infections and infestations) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Pneumonia (Infections and infestations) | 2/147 (2) | 3/149 (3) | 1/147 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 0/147 (0) | 0/149 (0) | 1/147 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Dehydration (Metabolism and nutrition disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/147 (0) | 2/149 (2) | 0/147 (0)
Lung carcinoma, cell type unspecified, Stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Hypoaesthesia (Nervous system disorders) | 1/147 (1) | 0/149 (0) | 0/147 (0)
Syncope (Nervous system disorders) | 1/147 (1) | 1/149 (1) | 0/147 (0)
Syncope vasovagal (Nervous system disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Bladder prolapse (Renal and urinary disorders) | 1/147 (1) | 0/149 (0) | 0/147 (0)
Renal failure acute (Renal and urinary disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5/147 (6) | 7/149 (7) | 4/147 (4)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1/147 (1) | 0/149 (0) | 0/147 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0/147 (0) | 1/149 (1) | 0/147 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Formoterol 12 Mcg 2x/Day | Arformoterol 15 Mcg 2x/Day | Arformoterol 25 Mcg 2x/Day
Anemia (Blood and lymphatic system disorders) | 0/147 (0) | 4/149 (4) | 1/147 (1)
Palpitations (Cardiac disorders) | 3/147 (4) | 1/149 (1) | 0/147 (0)
Ear Pain (Ear and labyrinth disorders) | 1/147 (1) | 0/149 (0) | 3/147 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 3/147 (3) | 1/149 (1) | 0/147 (0)
Constipation (Gastrointestinal disorders) | 4/147 (4) | 2/149 (2) | 4/147 (4)
Diarrhoea (Gastrointestinal disorders) | 2/147 (2) | 5/149 (5) | 2/147 (2)
Dry mouth (Gastrointestinal disorders) | 1/147 (1) | 1/149 (1) | 3/147 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3/147 (3) | 5/149 (5) | 1/147 (1)
Nausea (Gastrointestinal disorders) | 5/147 (5) | 2/149 (2) | 0/147 (0)
Fatigue (General disorders) | 3/147 (3) | 4/149 (4) | 1/147 (1)
Non-cardiac chest pain (General disorders) | 3/147 (5) | 0/149 (0) | 1/147 (1)
Pain (General disorders) | 0/147 (0) | 4/149 (4) | 0/147 (0)
Pyrexia (General disorders) | 1/147 (1) | 6/149 (6) | 3/147 (3)
Bronchitis (Infections and infestations) | 9/147 (11) | 8/149 (12) | 10/147 (12)
Diverticulitis (Infections and infestations) | 0/147 (0) | 4/149 (4) | 0/147 (0)
Influenza (Infections and infestations) | 3/147 (3) | 2/149 (2) | 1/147 (1)
Nasopharyngitis (Infections and infestations) | 17/147 (21) | 8/149 (10) | 15/147 (21)
Rhinitis (Infections and infestations) | 1/147 (1) | 3/149 (3) | 2/147 (2)
Sinusitis (Infections and infestations) | 4/147 (6) | 4/149 (4) | 7/147 (8)
Upper respiratory tract infection (Infections and infestations) | 6/147 (6) | 4/149 (6) | 6/147 (6)
Viral infection (Infections and infestations) | 1/147 (1) | 2/149 (2) | 4/147 (6)
Hypokalemia (Metabolism and nutrition disorders) | 3/147 (3) | 1/149 (1) | 1/147 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/147 (3) | 1/149 (1) | 2/147 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4/147 (4) | 3/149 (3) | 3/147 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6/147 (11) | 4/149 (5) | 7/147 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3/147 (3) | 1/149 (1) | 0/147 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/147 (8) | 2/149 (2) | 2/147 (3)
Dizziness (Musculoskeletal and connective tissue disorders) | 7/147 (8) | 3/149 (3) | 1/147 (1)
Headache (Musculoskeletal and connective tissue disorders) | 4/147 (6) | 6/149 (9) | 10/147 (12)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 22/147 (28) | 34/149 (45) | 35/147 (43)
Cough (Respiratory, thoracic and mediastinal disorders) | 2/147 (2) | 1/149 (1) | 4/147 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2/147 (2) | 4/149 (4) | 3/147 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/147 (2) | 2/149 (2) | 5/147 (5)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3/147 (3) | 1/149 (1) | 1/147 (1)
Hypertension (Vascular disorders) | 3/147 (3) | 3/149 (3) | 6/147 (6)
Urinary tract infection (Infections and infestations) | 5/147 (6) | 4/149 (6) | 5/147 (5)
Candidiasis (Infections and infestations) | 3/147 (4) | 1/149 (1) | 1/147 (1)
Ear Infection (Infections and infestations) | 0/147 (0) | 0/149 (0) | 3/147 (3)
Oral Pain (Gastrointestinal disorders) | 1/147 (1) | 1/149 (1) | 3/147 (3)

LIMITATIONS AND CAVEATS:
Please see dropout rate in participant group. Sunovion is unaware of any other limitations or caveats associated with this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.